CLINICAL TRIAL: NCT01496131
Title: A Randomized Phase II Study of Tecemotide in Combination With Standard Androgen Deprivation Therapy and Radiation Therapy for Untreated, Intermediate and High Risk Prostate Cancer Patients
Brief Title: Tecemotide (L-BLP25) in Prostate Cancer
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: EMD Serono (Industry)
Collaborators: National Cancer Institute (NCI) (NIH)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: EMR 63325-015; BB-IND 7787 (Other: CBER)
Record Dates: First submitted 2011-11-03; First posted 2011-12-21 (Estimated); Results first posted 2018-03-09 (Actual); Last update posted 2018-03-09 (Actual); Status verified 2018-02

CONDITIONS: Prostate Cancer
Keywords: Tecemotide; Prostate Cancer; Goserelin; Cyclophosphamide; Radiotherapy
MeSH Terms: conditions — Prostatic Neoplasms | interventions — Radiotherapy; Goserelin; Cyclophosphamide; L-BLP25

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Standard therapy (Active Comparator): Radiation therapy in combination with androgen deprivation therapy (ADT).
  Interventions: Radiation: Radiation therapy; Drug: Goserelin
- Standard therapy plus tecemotide (L-BLP25) (Experimental): Standard therapy (radiation therapy in combination with ADT) plus tecemotide (L-BLP25).
  Interventions: Radiation: Radiation therapy; Drug: Goserelin; Drug: Cyclophosphamide; Drug: Tecemotide (L-BLP25)

INTERVENTIONS:
Radiation: Radiation therapy — Radiation therapy will be administered at a daily dose of 180 centigrays (cGy) 5 days a week for approximately 6 to 8 weeks.
Drug: Goserelin — ADT (Goserelin) will be administered at a dose of 10.8 milligrams (mg) subcutaneously every 3 months for 24 months for the high risk group and for 6 months in the intermediate risk group, starting 2-3 months prior to radiation therapy.
Drug: Cyclophosphamide — Cyclophosphamide will be administered at a single dose of 300 milligrams per square meter (mg/m^2) to a maximum of 600 mg, as an intravenous injection 3 days prior to the first administration of tecemotide (L-BLP25).
  Arms: Standard therapy plus tecemotide (L-BLP25)
Drug: Tecemotide (L-BLP25) — Tecemotide (L-BLP25) will be administered at a dose of 918 microgram (mcg) as subcutaneous injection every 2 weeks for 5 doses followed by every 6 weeks for an additional 4 doses, starting 2-3 months prior to radiation therapy and on the same day that ADT began.
  Other Names: L-BLP25; BLP25 liposome vaccine; Epipepimut-S
  Arms: Standard therapy plus tecemotide (L-BLP25)

SUMMARY:
This study examines tecemotide (L-BLP25) in combination with standard treatment for prostate cancer.

ELIGIBILITY:
Inclusion Criteria:

* Histopathologic documentation of prostate cancer confirmed at the institution of study enrollment prior to starting this study
* Newly diagnosed or previously untreated prostate cancer with intermediate or high risk features as defined in the protocol
* No evidence of metastatic disease on computed tomography (CT) / magnetic resonance imaging (MRI) or bone scans
* No systemic steroid use within 2 weeks prior to initiation of experimental therapy. Limited doses of systemic steroids to prevent intravenous contrast, allergic reaction or anaphylaxis (in subjects who have known contrast allergies) are allowed
* Eastern Co-operative Oncology Group (ECOG) performance status of 0-1
* Human leukocyte antigen (HLA)-A2 or A3 positive for immunologic monitoring
* Hematological and biochemical eligibility parameters as defined in the protocol
* No other active malignancies within the past 3 years (with the exception of non-melanoma skin cancers or carcinoma in situ of the bladder)
* Willing to travel to the study center(s) for follow-up visits
* Age greater than or equal to 18 years old
* Able to understand and sign informed consent
* Must agree to use effective birth control (such as a condom) or abstinence during and for a period of 4 months after the last administration of immunotherapy

Exclusion Criteria:

* No evidence of being immunocompromised by human immunodeficiency virus, a medical condition requiring systemic steroids, a medical condition requiring immunosuppressive therapy, splenectomy
* Active Hepatitis B or Hepatitis C
* Subjects should have no autoimmune diseases that have required treatment as specified in the protocol
* History of immunodeficiency diseases, hereditary or congenital immunodeficiencies
* Serious intercurrent medical illness
* A clinically significant cardiac disease
* Subjects who have received any prior therapy for prostate cancer
* Subjects who have known brain metastasis, or with a history of seizures, encephalitis, or multiple sclerosis
* Subjects receiving any other investigational agents
* Contraindication to biopsy such as bleeding disorders, ratio of prothrombin time to partial thromboplastin time (PT/PTT) >=1.5 times the upper limit of normal, artificial heart valve
* Contraindication to MRI such as subjects weighing >136 kilograms, allergy to magnetic resonance (MR) contrast agent, subjects with pacemakers, cerebral aneurysm clips, shrapnel injury or implantable electronic devices
* Contraindication to radiation therapy such as pre-existing and active prostatitis or proctitis, inflammatory bowel disease or known genetic sensitivity to ionizing radiation, or history of prior radiation to the pelvis

Min Age: 18 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 28 (Actual)
Dates: Start 2011-10-24 (Actual); Primary Completion 2016-11-25 (Actual); Study Completion 2016-11-25 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Medical Responsible, Study Director — EMD Serono, an affiliate of MerckKGaA, Darmstadt, Germany
Locations (1):
- Please Contact US Medical Information, Rockland, Massachusetts, United States

RESULTS

PARTICIPANT FLOW:
Recruitment Details: First subject First Visit/Last Subject Last Visit: 24 October 2011/25 November 2016.
Groups:
- Standard Therapy: Subjects received Goserelin 10.8 milligrams (mg) subcutaneously every 3 months for 2 years and radiation therapy lasting 6-8 weeks starting 2-3 months after Androgen Deprivation Therapy (ADT).
- Standard Therapy Plus Tecemotide (L-BLP25): Subjects received Goserelin 10.8 mg subcutaneously every 3 months for 2 years and radiation therapy lasting 6-8 weeks starting 2-3 months after ADT. In addition to the above standard treatment, subjects received tecemotide at a dose of 918 microgram (mcg) as subcutaneous injections every 2 weeks for 2 months followed by continuation treatment with 4 doses of tecemotide every 6 weeks. Subjects also received a single dose of cyclophosphamide 300 mg per square meter intra-venously 3 days before 1st administration of tecemotide.
Period: Overall Study
Arm/Group | Standard Therapy | Standard Therapy Plus Tecemotide (L-BLP25)
Started | 14 | 14
Completed | 14 | 14
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Population: Baseline population included all randomized subjects.
Units Other Than Participants: Subjects
Groups:
- Standard Therapy: Subjects received Goserelin 10.8 milligrams (mg) subcutaneously every 3 months for 2 years and radiation therapy lasting 6-8 weeks starting 2-3 months after ADT.
- Total: Total of all reporting groups
Arm/Group | Standard Therapy | Standard Therapy Plus Tecemotide (L-BLP25) | Total
Number analyzed (Participants) | 14 | 14 | 28
Number analyzed (Subjects) | 14 | 14 | 28
Age, Continuous [Median (Full Range); unit: years] | 69.0 [48 to 75] | 64 [54 to 78] | 64.5 [48 to 78]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 0 | 0 | 0
  Male | 14 | 14 | 28

OUTCOME MEASURES:

1. Primary Outcome: Number of Subjects With Change From Baseline in the Mucinous Glycoprotein 1 (MUC1) Specific Systemic T-Cells Immune Response at Day 60 (Pre-Radiation)
Description: MUC1-specific systemic immune response was measured by intracellular cytokine antigen specific staining following a period of in vitro stimulation (IVS) with overlapping 15-mer peptide pools encoding the tumor-associated antigen (TAA) MUC-1. Baseline was defined as the measurement taken prior to the first dose of study medication (Day 1).
Time Frame: Baseline and Day 60 (Pre-Radiation)
Population: Analysis population included only subjects who had scored positive to viral pool in peripheral blood mononuclear cells and were considered as evaluable. Here, "Number of Participants Analyzed" signifies subjects evaluable for this outcome measure.
Measure: Count of Participants; unit: Participants
Arm/Group | Standard Therapy | Standard Therapy Plus Tecemotide (L-BLP25)
Number analyzed (Participants) | 9 | 8
Participants | 2 | 3

2. Primary Outcome: Number of Subjects With Change From Baseline in the Mucinous Glycoprotein 1 (MUC1) Specific Systemic T-Cells Immune Response at Day 190 (Post-radiation)
Description: as for outcome 1
Time Frame: Baseline and Day 190 (Post-radiation)
Population: as for outcome 1
Measure: Count of Participants; unit: Participants
Arm/Group | Standard Therapy | Standard Therapy Plus Tecemotide (L-BLP25)
Number analyzed (Participants) | 8 | 6
Participants | 1 | 1

3. Secondary Outcome: Number of Subjects With Progression/Recurrence Status Based on Prostate-specific Antigen (PSA) Levels
Description: Progression/recurrence status was reported based on Prostate-specific Antigen (PSA) Levels. Recurrence of PSA after completion of therapy represents disease progression and was determined using the American Society for Therapeutic Radiology and Oncology (ASTRO) "Phoenix criteria". These criteria define biochemical recurrence after radiation therapy as a PSA level equal to the lowest (nadir) PSA level achieved after therapy plus 2 nanogram per milliliter.
Time Frame: From randomization up to 24 months
Population: Analysis population included all subjects randomized in the study.
Measure: Count of Participants; unit: Participants
Arm/Group | Standard Therapy | Standard Therapy Plus Tecemotide (L-BLP25)
Number analyzed (Participants) | 14 | 14
Participants | 2 | 0

4. Secondary Outcome: Number of Subjects With a Doubling in Number of T-cells in Tumor Biopsy From Baseline at Pre-radiotherapy (Pre-RT) and Post-radiotherapy (Post-RT)
Description: Doubling in number of T-cells was assessed by immunologic responses (in the tumor microenvironment) in subjects consenting to undergo study biopsies. Baseline was defined as the measurement taken within 8 weeks of prior to the first dose of study medication (Day 1).
Time Frame: Baseline, Week 6-12 (Pre-RT), Week 40 (Post-RT)
Population: Analysis population included only the subjects who were randomized and provided consent for biopsy and whose baseline measurement was considered as evaluable. Here, "number analyzed" signifies subjects evaluable at specified time point and "number analyzed"=0 signifies that no subjects were evaluable at the specified time point.
Measure: Count of Participants; unit: Participants
Arm/Group | Standard Therapy | Standard Therapy Plus Tecemotide (L-BLP25)
Number analyzed (Participants) | 1 | 7
Participants
  Pre-RT: number analyzed (Participants) | 1 | 2
  Pre-RT | 1 | 1
  Post-RT: number analyzed (Participants) | 0 | 1
  Post-RT |  | 1

ADVERSE EVENTS:
Arm/Group | Standard Therapy | Standard Therapy Plus Tecemotide (L-BLP25)
All-Cause Mortality (participants affected / at risk) | 0/14 | 0/14
Serious Adverse Events (participants affected / at risk) | 1/14 | 2/14
Other Adverse Events (participants affected / at risk) | 14/14 | 14/14
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Standard Therapy (N=14) | Standard Therapy Plus Tecemotide (L-BLP25) (N=14)
Abdominal pain (Gastrointestinal disorders) | 0 | 1
Diarrhoea (Gastrointestinal disorders) | 0 | 1
Crohn's disease (Gastrointestinal disorders) | 0 | 1
Small intestinal obstruction (Gastrointestinal disorders) | 0 | 1
Osteoarthritis;hip replacement surgery (Musculoskeletal and connective tissue disorders) | 0 | 1
Lumbar stenosis (Musculoskeletal and connective tissue disorders) | 0 | 1
Presyncope (Nervous system disorders) | 1 | 0
Ileocecectomy and resection (Surgical and medical procedures) | 0 | 1
Laminectomy (Surgical and medical procedures) | 0 | 1
Hypotension (Vascular disorders) | 1 | 0
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Standard Therapy (N=14) | Standard Therapy Plus Tecemotide (L-BLP25) (N=14)
Anaemia (Blood and lymphatic system disorders) | 7 | 9
Atrioventricular block first degree (Cardiac disorders) | 0 | 1
Palpitations (Cardiac disorders) | 1 | 0
Vertigo (Eye disorders) | 1 | 0
Eye Redness and discomfort in left Eye (Eye disorders) | 0 | 1
Vision blurred (Eye disorders) | 1 | 0
Sinus tachycardia (Cardiac disorders) | 1 | 0
Abdominal distension (Gastrointestinal disorders) | 0 | 1
Abdominal pain (Gastrointestinal disorders) | 0 | 2
Anal incontinence (Gastrointestinal disorders) | 1 | 0
Constipation (Gastrointestinal disorders) | 0 | 3
Diarrhoea (Gastrointestinal disorders) | 4 | 7
Dry mouth (Gastrointestinal disorders) | 0 | 1
Flatulence (Gastrointestinal disorders) | 0 | 2
GI bleed - GI Virus (Gastrointestinal disorders) | 1 | 0
Gastrooesophageal reflux disease (Gastrointestinal disorders) | 1 | 0
Haemorrhoidal haemorrhage (Gastrointestinal disorders) | 0 | 1
Haemorrhoids (Gastrointestinal disorders) | 2 | 1
Nausea (Gastrointestinal disorders) | 1 | 3
Proctalgia (Gastrointestinal disorders) | 0 | 1
Proctitis (Gastrointestinal disorders) | 3 | 0
Rectal haemorrhage (Gastrointestinal disorders) | 1 | 0
Vomiting (Gastrointestinal disorders) | 0 | 1
Chills (General disorders) | 1 | 0
Fatigue (General disorders) | 10 | 11
Influenza like illness (General disorders) | 0 | 1
Injection site reaction (General disorders) | 1 | 10
Non-cardiac chest pain (General disorders) | 1 | 0
Oedema peripheral (General disorders) | 2 | 3
Pain (General disorders) | 1 | 3
Pyrexia (General disorders) | 1 | 0
Scabies (Infections and infestations) | 0 | 1
Skin infection (Infections and infestations) | 1 | 0
Upper respiratory tract infection (Infections and infestations) | 1 | 1
Contusion (Injury, poisoning and procedural complications) | 1 | 0
Fall (Injury, poisoning and procedural complications) | 1 | 0
Fracture (Injury, poisoning and procedural complications) | 0 | 1
Recall phenomenon (Injury, poisoning and procedural complications) | 1 | 0
Alanine aminotransferase increased (Investigations) | 0 | 6
Aspartate aminotransferase increased (Investigations) | 0 | 3
Blood alkaline phosphatase increased (Investigations) | 1 | 1
Blood creatine phosphokinase increased (Investigations) | 0 | 2
Blood creatinine increased (Investigations) | 1 | 3
CD4 lymphocytes decreased (Investigations) | 9 | 13
Lymphocyte count decreased (Investigations) | 12 | 14
Neutrophil count decreased (Investigations) | 3 | 3
Platelet count decreased (Investigations) | 0 | 5
Weight increased (Investigations) | 0 | 1
White blood cell count decreased (Investigations) | 9 | 7
Decreased appetite (Metabolism and nutrition disorders) | 0 | 2
Hypercalcaemia (Metabolism and nutrition disorders) | 0 | 3
Hyperglycaemia (Metabolism and nutrition disorders) | 8 | 10
Hyperkalaemia (Metabolism and nutrition disorders) | 1 | 3
Hypermagnesaemia (Metabolism and nutrition disorders) | 0 | 1
Hypernatraemia (Metabolism and nutrition disorders) | 4 | 4
Hypoalbuminaemia (Metabolism and nutrition disorders) | 1 | 3
Hypoglycaemia (Metabolism and nutrition disorders) | 2 | 0
Hypokalaemia (Metabolism and nutrition disorders) | 1 | 0
Hypomagnesaemia (Metabolism and nutrition disorders) | 1 | 2
Hyponatraemia (Metabolism and nutrition disorders) | 0 | 1
Hypophosphataemia (Metabolism and nutrition disorders) | 1 | 1
Polydipsia (Metabolism and nutrition disorders) | 1 | 0
Arthralgia (Musculoskeletal and connective tissue disorders) | 0 | 1
Arthritis (Musculoskeletal and connective tissue disorders) | 0 | 1
Back pain (Musculoskeletal and connective tissue disorders) | 0 | 1
Muscular weakness (Musculoskeletal and connective tissue disorders) | 1 | 0
Myalgia (Musculoskeletal and connective tissue disorders) | 0 | 3
Pain in extremity (Musculoskeletal and connective tissue disorders) | 4 | 1
Dizziness (Nervous system disorders) | 2 | 0
Dysgeusia (Nervous system disorders) | 1 | 0
Headache (Nervous system disorders) | 1 | 1
Peripheral sensory neuropathy (Nervous system disorders) | 1 | 2
Anxiety (Psychiatric disorders) | 1 | 0
Insomnia (Psychiatric disorders) | 1 | 0
Hesitancy (Psychiatric disorders) | 1 | 0
Cystitis noninfective (Renal and urinary disorders) | 2 | 4
Haematuria (Renal and urinary disorders) | 2 | 2
Haemoglobinuria (Renal and urinary disorders) | 0 | 1
Micturition urgency (Renal and urinary disorders) | 1 | 1
Pollakiuria (Renal and urinary disorders) | 3 | 0
Proteinuria (Renal and urinary disorders) | 0 | 1
Urinary incontinence (Renal and urinary disorders) | 1 | 1
Breast pain (Reproductive system and breast disorders) | 0 | 1
Erectile dysfunction (Reproductive system and breast disorders) | 3 | 1
Gynaecomastia (Reproductive system and breast disorders) | 1 | 1
Scrotal pain (Reproductive system and breast disorders) | 1 | 0
Cough (Respiratory, thoracic and mediastinal disorders) | 2 | 0
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 1 | 1
Oropharyngeal pain (Respiratory, thoracic and mediastinal disorders) | 0 | 1
Dermatitis acneiform (Skin and subcutaneous tissue disorders) | 1 | 0
Dry skin (Skin and subcutaneous tissue disorders) | 1 | 1
Rash maculo-papular (Skin and subcutaneous tissue disorders) | 1 | 0
Tick bite (Skin and subcutaneous tissue disorders) | 0 | 1
Skin induration (Skin and subcutaneous tissue disorders) | 0 | 1
Hot flush (Vascular disorders) | 13 | 11
Hypertension (Vascular disorders) | 0 | 2
Hypotension (Vascular disorders) | 1 | 0
Early satiety (Metabolism and nutrition disorders) | 0 | 1

LIMITATIONS AND CAVEATS:
For primary outcome measure, antigen specific data was provided with updated technique. Enzyme-Linked ImmunoSpot technique was not done, but intracellular cytokine antigen specific responses was evaluated, which is now the lab technique used.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No